CLINICAL TRIAL: NCT04057625
Title: Transthoracic Ultrasound in the Diagnosis and Follow-up of Ventilator Associated Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, dina reda ragab gharieb, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: sonar in vap
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Ventilator Associated Pneumonia; Lung Ultrasound
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung ultrasound (Other): using lung ultrasound in diagnosis and follow up of vap measuring the largest area of consolidation according to intercostal space and the direction of the probe
  Interventions: Device: transthoracic ultrasound

INTERVENTIONS:
Device: transthoracic ultrasound — using transthoracic ultrasound in the diagnosis and follow up of vap,measuring the largest area of consolidation according to intercostal space and the direction of the probe.

SUMMARY:
To evaluate the sensitivity, specificity and diagnostic accuracy of bedside transthoracic ultrasound examination in the diagnosis and follow up of ventilator associated pneumonia.

DETAILED DESCRIPTION:
VAP is the most frequent hospital-acquired infection in intensive care units. Depending on the diagnostic criteria used, its incidence ranges from 5% to 67%. The risk of acquiring VAP is 3% per day during the first 5 days on mechanical ventilation, and it is decreased to 1% per day for the following days.

VAP is suspected when subject shows high grade fever, increase in leukocyte count, change in color of sputum and tachypnea. It's a leading cause of mortality in 15- 65% of the cases.

Serial chest x-ray for diagnosis and follow up, done at time of diagnosis, after 5 days and after 10 days. Chest radiography is consistently carried out after LUS , LUS is done every other day, measuring the largest area of consolidation according to the intercostal space and direction of the probe . Chest radiography is read by two physicians.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for at least 48 hours.
* New or evolving infiltrate on chest radiograph (CXR).
* Clinical pulmonary infection score more than or equal 6

Exclusion Criteria:

* Patients who are less than 18 years old.
* Patients who have evidence of pneumonia before or prior to being mechanically ventilated.
* Patients with pulmonary infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
detecting ultrasound efficiency in diagnosis and follow up of vap | baseline
  Sensitivity, specificity, and diagnostic accuracy of lung ultrasound to diagnose and follow up ventilator-associated pneumonia.

SECONDARY OUTCOMES:
icu stay | baseline
  Duration of stay in ICU.
hospital stay | basline
  Duration of hospital stay.
mortality | basline
  mortality from vap

IPD SHARING:
Plan to Share IPD: Yes